CLINICAL TRIAL: NCT02838186
Title: Diagnostic Yield of Scope Retroflexion in the Right Colon: A Prospective Cohort Study
Brief Title: Backwards Examination of the Right Colon: A Back-to-back Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, ATHANASIOS SIOULAS, Dr., Attikon Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Retro-2013
Record Dates: First submitted 2013-06-19; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Colon Neoplasms
Keywords: colonoscopy; right colon retroflexion; adenoma detection rate; feasibility; surveillance interval
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- right colon in retroflexion (Active Comparator): * polyp/adenoma detection
  * feasibility
  Interventions: Procedure: retroflexion
- right colon in forward view (Active Comparator): polyp/adenoma detection
  Interventions: Procedure: forward view

INTERVENTIONS:
Procedure: retroflexion — examination of the right colon with scope retroflexion
  Arms: right colon in retroflexion
Procedure: forward view — examination of the right colon in forward view
  Arms: right colon in forward view

SUMMARY:
The aim of this study is to evaluate the examination of the proximal colon with the retroflexion colonoscopic technique in terms of feasibility and its possible additive contribution in the detection of important lesions, namely polyps and cancers.

DETAILED DESCRIPTION:
The investigators prospectively examined the additional diagnostic yield of right colon examination with colonoscope retroflexion in consecutive, symptomatic and screening - surveillance patients. Right colon was examined in forward-view first and thereafter, retroflexion was performed to re-inspect it.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective colonoscopy in a Attikon University General Hospital.

Exclusion Criteria:

* patients aged <18 and >80 years;
* right colectomy;
* recent abdominalsurgery;
* multiple diverticula of the right colon;
* American Society of Anesthesiology (ASA) physical status classification grade IV;
* inflammatory bowel disease and polyposis syndromes.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
number of additional identified polyps with right colon scope retroflexion | one week

SECONDARY OUTCOMES:
Change in colorectal cancer (CRC) surveillance intervals among screening-surveillance patients | one week
  change: YES or NO
Rate of retroflexion-related adverse events. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Triantafyllou, Prof, Study Director — Hepatogastroenterology Unit, 2nd Department of Internal Medicine and Research Institute, Attikon University General Hospital, University of Athens, Greece
Locations (1):
- Attikon University General Hospital, Haidari, Attica, Greece

REFERENCES:
- [Background] van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systematic review. Am J Gastroenterol. 2006 Feb;101(2):343-50. doi: 10.1111/j.1572-0241.2006.00390.x. PMID 16454841
- [Background] Vemulapalli KC, Rex DK. Evolving techniques in colonoscopy. Curr Opin Gastroenterol. 2011 Sep;27(5):430-8. doi: 10.1097/MOG.0b013e328349cfc0. PMID 21785352